CLINICAL TRIAL: NCT05083117
Title: Safety and Efficacy of Inhaled XW001 (Interleukin 29 Analog for Nebulization) For Hospitalized COVID-19 Patients Requiring Oxygen Therapy: A Multiregional, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Safety and Efficacy of Inhaled XW001 For Hospitalized COVID-19 Patients Requiring Oxygen Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in COVID-19 subject enrollment
Sponsor: Sciwind Biosciences APAC CO Pty. Ltd. (Industry)
Collaborators: Sciwind Biosciences USA Co., Ltd. (Industry); Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCW1201-3121
Record Dates: First submitted 2021-10-17; First posted 2021-10-19 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — XW001

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XW001 (Experimental): Treatment arm patients will receive inhaled XW001 1 mg, once daily, using a commercially available nebulizer (Aerogen Solo, Aerogen Ireland) for up to 14 days. Treatment should be continued until discharge or progression to score 6 or higher but maximum up to 14 days. Dosing must be started within 48 hours of hospitalization.
  Interventions: Drug: XW001
- Placebo (Placebo Comparator): Placebo arm patients will receive volume-matching placebo 1 mL, once daily, using a commercially available nebulizer (Aerogen Solo, Aerogen Ireland) for up to 14 days. Treatment should be continued until discharge or progression to score 6 or higher but maximum up to 14 days. Dosing must be started within 48 hours of hospitalization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XW001 — It is anticipated that inhalation of 1 mg XW001 solution up to 14 days will result in a relatively lower systemic exposure in COVID-19 patients on oxygen therapy compared to that in healthy participants as COVID-19 patients tend to have impaired lung function of diffusive, restrictive, obstructive, or mixed origins.
  Other Names: IL-29 analog
  Arms: XW001
Drug: Placebo — It is anticipated that inhalation of 1 mg Placebo solution up to 14 days will result in a relatively lower systemic exposure in COVID-19 patients on oxygen therapy compared to that in healthy participants as COVID-19 patients tend to have impaired lung function of diffusive, restrictive, obstructive, or mixed origins.
  Arms: Placebo

SUMMARY:
This is a multiregional, randomized, double-blind, placebo-controlled Phase 2 study in patients with confirmed symptomatic COVID-19, designed to evaluate the safety, tolerability, efficacy, and PK of XW001 (IL-29 analog) inhalation solution. The purpose of this study is to evaluate whether treatment with XW001 reduces the likelihood of worsening disease in patients with severe COVID-19. Hospitalized patients on oxygen therapy by mask or nasal prongs (WHO-OSCI score 4) will be enrolled.

DETAILED DESCRIPTION:
Treatment arm patients will receive inhaled XW001 1 mg and placebo arm patients will receive volume-matching placebo 1 mL, once daily, using a commercially available nebulizer for up to 14 days. Treatment should be continued until discharge or progression to score 6 or higher but maximum up to 14 days. Dosing must be started within 48 hours of hospitalization. In addition, both the treatment groups will receive SoC.

The present study is a pilot in the development phase and comprising approximately 120 patients. An independent, external Data Monitoring Committee (DMC) will review all the preliminary clinical data available, including safety, tolerability, efficacy, and PK for the first 20 patients. The decision to recruit the subsequent 100 patients will solely depend on safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant or nonlactating female, aged 18 to 70 years at the time of consenting
2. Hospitalized due to infection with SARS-CoV-2 confirmed on validated local RT-PCR or other equivalent assays within 48 hours prior to screening and within 96 hours prior to randomization
3. Assessed to be hospitalized cases (rated at WHO-OSCI score 4 [on oxygen therapy by mask or nasal prongs]) within 24 hours prior to randomization
4. Admitted to hospital as clinically indicated for management of severe COVID-19 defined by the following criteria:

   * Positive RT-PCR test for SARS-CoV-2 or an equivalent test
   * Symptom suggestive of severe systemic illness with COVID-19, which could include any symptom of moderate illness or shortness of breath at rest, or respiratory distress
   * Clinical signs indicative of severe illness with COVID-19, being given oxygenation and meeting one of the following:

     * Respiratory rate ≥30 breaths per minute
     * Heart rate ≥125 beats per minute
     * Oxygen saturation (SpO2) <94% on room air at sea level
     * Arterial partial pressure of oxygen (PaO2)/fraction of inspired oxygen (FiO2) <300 mmHg or SpO2/FiO2 <315 mmHg
     * Lung infiltrates >50%
   * No criteria for critical severity
5. Female of childbearing potential must be postmenopausal for 1 year or longer, surgically sterile or having used a medically effective method of contraception for at least 3 months prior to hospitalization
6. Willing and able to provide a signed and dated or electronic informed consent for participation in this study.

Exclusion Criteria:

Patients will be excluded from the study if they satisfy any of the following criteria at the screening visit unless otherwise stated:

1. Having become symptomatic (fever, cough, and other likely symptoms) or positive on virologic test for more than 8 days prior to hospitalization
2. Diagnosed with SARS-CoV-2 confirmed more than 48 hours prior to hospitalization, otherwise reconfirmed positive on repeated RT-PCR (local laboratory) or other equivalent assays within 48 hours prior to randomization
3. Having been hospitalized for more than 48 hours, or showing a worsening medical condition within 48 hours after hospitalization in the opinion of the investigator
4. Known to have received any approved or investigational COVID-19 vaccines within 6 months prior to randomization. Vaccination records can be self-reported by the patient if there is no recorded history
5. Known to have received any approved or investigational therapeutic agents against SARS-CoV-2 including convalescent plasma, monoclonal antibodies, except for remdesivir, dexamethasone, or IL-6 inhibitors as a part of SoC
6. Having received any investigational medicinal products within 90 days of randomization
7. On noninvasive ventilation, eg, continuous positive airway pressure or bilevel positive airway pressure or high-flow oxygen therapy (at WHO-OSCI score 5)
8. Intubated, ventilated (invasively), on any advanced organ/life support (pressors, renal replacement therapy, ECMO), or remaining in the intensive care unit (at WHO-OSCI score 6 and 7)
9. Known to be hypersensitive or allergic to any natural or recombinant protein products
10. Inability to utilize nebulized drugs, or history of bronchospasm with inhaled medications
11. Patients with cardiac disease (New York Heart Association III/IV), liver cirrhosis (>5 x upper limit of normal [ULN]), on chemotherapy, dialysis patients with estimated glomerular filtration rate <30 mL/min/1.73m2, or have other debilitating condition or any other clinically significant medical condition or laboratory abnormality that, in the opinion of the investigator, would jeopardize the safety of the patient or non- COVID-19 irreversible underlying condition with projected fatal course within 6 months or with high-risk of mortality
12. Female patients are pregnant or lactating, or male or female patients have a childbearing plan within 30 days prior to randomization until 90 days after the last dosing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-30 (Estimated); Primary Completion 2022-03-10 (Estimated); Study Completion 2022-04-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | 35 days
  Incidence of treatment-emergent adverse events (TEAEs), grade ≥3 TEAEs, SAEs, TEAEs leading to premature discontinuation of study treatment, TEAEs leading to study discontinuation, and TEAEs leading to deaths
Change from the baseline in clinical laboratory results | 35 days
  Percentage of the lab results change
Incidence of clinically significant laboratory findings | 35 days
  Percentage of the lab results change
Change from the baseline in vital signs results | 35 days
  Vital signs will be recorded twice daily while the patient is hospitalized. Vital signs may also be performed at other times if judged clinically appropriate or if the ongoing review of the data suggests a more detailed assessment of vital signs is required.
Change from the baseline in electrocardiogram (ECG) findings | 35 days
  A 12-lead ECG is to be performed at screening in the supine position and at rest for at least 5 minutes. Additionally, a 12-lead ECG will be performed if QT abnormality is noted or early termination while the patient is hospitalized or at the discretion of the investigator.

SECONDARY OUTCOMES:
Time to clinical improvement from the time of randomization. | 28 days
  Time to clinical improvement is defined as the time (in days) from the randomization date to the first day on which a patient satisfies a score of 0, 1, 2, or 3 on the 9-point WHO-OSCI and maintains a score ≤3 at least 48 hours (initial improvement) and maintains this up to the 28-day timeframe (sustained improvement)
Time to hospital discharge from the time of randomization | 28 days
  At or below WHO-OSCI score 2 from the time of randomization
Time to clinical recovery from the time of randomization | 28 days
  Time of clinical recovery (in days) will be calculated using the WHO-OSCI from the randomization date to the first day on which the patient satisfies a score of 0 or 1 on the 9-point WHO-OSCI and remains at 0 or 1 until Day 28 (has no subsequent readmission for COVID-19 signs or symptoms)
Time to viral clearance | 28 days
  targeted not detected on real-time quantitative polymerase chain reaction [qPCR] assay) from the time of randomization
Viral load kinetics on real-time qPCR assay | 28 days
  A real-time qPCR will be done to determine the viral load kinetics in positive RT-PCR samples.
Proportions of patients experiencing clinical improvement, hospital discharge, clinical recovery, and viral clearance | 28 days
  The proportions of patients will be compared using the logistic regression.
Proportion of patients experiencing clinical progression from the time of randomization | 35 days
  The proportions of patients will be compared using the logistic regression.
Proportion of patients progressing to on noninvasive ventilation or high-flow oxygen from the time of randomization | 35 days
  The proportions of patients will be compared using the logistic regression.
Proportion of patients progressing to on intubation with ventilation from the time of randomization | 35 days
  The proportions of patients will be compared using the logistic regression.
Proportion of patients progressing to death from the time of randomization | 35 days
  Proportion of patients progressing to death (WHO-OSCI score 8) within the 35-day timeframe from the time of randomization
Changes from the baseline in the BCSS total score and breathlessness and cough subscores | 35 days
  Change from the baseline in the BCSS scores will also be evaluated daily. A physical examination including height and weight will be measured. Height will be measured at screening only. If a patient is not able to stand easily, the patient may provide height.
Changes from the baseline in the NEWS2 | 35 days
  Change from the baseline in the NEWS2 scores will also be evaluated daily. A physical examination including height and weight will be measured. Height will be measured at screening only. If a patient is not able to stand easily, the patient may provide height.

OTHER OUTCOMES:
Serum XW001 concentration and appropriate serum XW001 | 35 days
  PK parameters determined via the noncompartmental analysis (intensive PK cohort only) or a population PK analysis approach
Proportions of patients with newly emerging serum anti-XW001 antibody | 35 days
  Proportions of anti-XW001 antibody after the randomization compared to the baseline (at the time of randomization).

CONTACTS AND LOCATIONS:
Overall Officials: Eddie Angles, Principal Investigator — Hospital Nacional Arzobispo Loayza; Ricardo Teijeiro, Principal Investigator — Hospital Pirovano
Locations (2):
- Hospital Pirovano, CABA, Bs AS, Argentina
- Hospital Nacional Arzobispo Loayza, Lima, Peru

IPD SHARING:
Plan to Share IPD: No